CLINICAL TRIAL: NCT02533635
Title: Product Functional Study of Effect A Master Ganoderma Detox Tea on Eczema Patient
Brief Title: Ganoderma Tea on Eczema Patient
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Principal Investigator, Shi Ping Zhang, Associate Professor, Hong Kong Baptist University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HongKongBU
Record Dates: First submitted 2015-08-18; First posted 2015-08-27 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Eczema
MeSH Terms: conditions — Eczema

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A-first intervention (Experimental): Subjects in Arm A receive Ganoderma tea (30g) daily for 8 weeks initially, followed by 8 weeks no intervention.
  Interventions: Dietary Supplement: A Master Ganoderma Detox Tea
- B-second intervention (Experimental): Subjects in Arm B receive no intervention for 8 weeks initially, followed by receiving Ganoderma tea (30g) daily for 8 weeks .
  Interventions: Dietary Supplement: A Master Ganoderma Detox Tea

INTERVENTIONS:
Dietary Supplement: A Master Ganoderma Detox Tea — A Master Ganoderma Detox Tea is consisted of GANODERMA, HERBA HOUTTUYNIAE, GLYCYRRHIZAE RADIX ET RHIZOMA and RUCTUS MOMORDICAE.
  Other Names: 老和尚靈芝健康茶（又名老和尚靈芝排毒茶）

SUMMARY:
This is a single-blind, cross-over pilot study to observe the safety and efficacy of Ganoderma tea on eczema patients.

DETAILED DESCRIPTION:
Objective This study is to conduct a preliminary observation on the effect of A Master Ganoderma Detox Tea in improving eczema symptoms. Because it is a preliminary study, there will not be a placebo control. However, in order to exclude the impact of spontaneous improvement, we will set up a cross over control group. Thus, we want to find out whether there is any difference in taking the tea and without taking the tea.

Research Design This is a randomized, cross-over-control and assessor-blinded clinical trial. Subjects will be divided into groups A and group B. Group A will receive the intervention for 8 weeks, followed by an 8-week period of no intervention. Group B will be observed without having any intervention for 8 weeks, and then receive the intervention for 8 weeks. Randomization will be carried out using a computer program.

Interventions Subjects in the treatment group (A) will take the A Master Ganoderma Detox Tea for 8 weeks. Initially, the dosage is twice a day, one pack (5g) each time, and then increased to three times a day, two packs each time within two weeks. The control group (B) will not receive any study intervention for 8 weeks, followed by similar intervention for 8 weeks.

In case of allergies or severe adverse reactions occur, the subject should stop taking the tea immediately and be excluded from the trial. During the control or intervention period, if necessary, subject may use short-term steroids or other topical medication to relieve the symptoms of eczema.

ELIGIBILITY:
Inclusion Criteria:

* eczema for 1 year, without other systemic illness.

Exclusion Criteria:

* severe systemic illness,
* oral steroid in the last month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-03 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Patient Oriented Eczema Measure | 16 weeks

SECONDARY OUTCOMES:
Eczema Area and Severity Index | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shi Ping Zhang, PhD, Principal Investigator — Hong Kong Baptist University
Locations (1):
- School of Chinese Medicine Building, Kowloon Tong, Kowloon, Hong Kong